CLINICAL TRIAL: NCT05638243
Title: Evaluation of a Model for the Early Diagnosis of Colorectal Cancer by the Detection of 5-hydroxymethylcytosine (5-hmC) in Plasma Cell-free DNA to the Community Colorectal Cancer Screening Program in Xuhui District, Shanghai
Brief Title: Evaluation of a Model for the Early Diagnosis of Colorectal Cancer by the Detection of 5-hydroxymethylcytosine (5-hmC) in Plasma Cell-free DNA to the Community Colorectal Cancer Screening Program
Acronym: METHOD-3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Director of Colorectal Surgery, Fudan University
Other Study IDs: METHOD-3
Record Dates: First submitted 2022-11-26; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High-risk residents

SUMMARY:
The incidence rate and mortality of colorectal cancer are increasing year by year. Most colorectal cancer develops from colorectal adenoma and is a disease that can be prevented and controlled. Thanks to early screening, the incidence rate and mortality of colorectal cancer have declined year by year. However, due to poor compliance with colonoscopy and the lack of efficient and convenient early screening methods, it is difficult to screen for colorectal cancer in China. According to the data from Shanghai Xuhui District Center for Disease Control and Prevention, the proportion of colonoscopies in high-risk groups for colorectal cancer is less than 18%.

This project plans to use the latest colorectal cancer screening technology, namely, 5hmC detection in peripheral blood and DNA methylation detection in feces, for those who are positive in the colorectal cancer incidence risk questionnaire or fecal occult blood in Xuhui District, Shanghai. It is strongly recommended that subjects with positive screening should undergo colonoscopy, to effectively improve the rate of colonoscopy and the early diagnosis rate of colorectal cancer. At the same time, to explore the screening efficiency of the early diagnosis model of 5hmC cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years old and<75 years old;

  * The initial screening was positive (fecal occult blood or colorectal cancer risk questionnaire was positive)； ③ Receive sample collection; ④ Sign the informed consent form.

Exclusion Criteria:

① History of colorectal cancer, colorectal adenoma, and treatment;

* Enteroscopy was performed after the initial screening was positive; ③ The subject or family members could not understand the conditions and objectives of the study or refused to participate in the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Xuhui District, Shanghai, who are initially screened as high-risk for colorectal cancer by Shanghai Xuhui District Center for Disease Control and Prevention, and do not receive a colonoscopy. People who are willing to accept the screening program.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects receiving colonoscopy | Three years
  Proportion of subjects receiving colonoscopy
Proportion of subjects suffering early colorectal cancer | Three years
  Proportion of stageⅠcancer in total colorectal cancer
Sensitivity and specificity of the model in the diagnosis of colorectal cancer and adenoma | Three years
  Sensitivity and specificity of the model in the diagnosis of colorectal cancer and adenoma

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, M.D.， PhD, Principal Investigator — Fudan University
Locations (1):
- Community Health Centers in Xuhui District, Shanghai, Shanghai Municipality, China